CLINICAL TRIAL: NCT04667247
Title: Multicenter Double Blind, Placebo Controlled RCT of Fomitopsis Officinalis and Trametes Versicolor to Treat COVID-19
Brief Title: RCT of Fomitopsis Officinalis and Trametes Versicolor to Treat COVID-19
Acronym: MACH19
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gordon Saxe (Other)
Collaborators: University of California, Los Angeles (Other); University of California, Irvine (Other)
Responsible Party: Sponsor-Investigator, Gordon Saxe, Director, Krupp Center for Integrative Research, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 200633-1a
Record Dates: First submitted 2020-12-03; First posted 2020-12-14 (Actual); Results first posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mushrooms (Experimental): Fomitopsis officinalis and Trametes versicolor
  Interventions: Drug: FoTv
- Placebo (Placebo Comparator): Organic brown rice
  Interventions: Drug: FoTv

INTERVENTIONS:
Drug: FoTv — 8 capsules three times a day for 14 consecutive days.
  Other Names: Fomitopsis officinalis and Trametes versicolor

SUMMARY:
This is a multi-center, randomized, double-blind, placebo-controlled clinical trial to evaluate two polypore mushrooms, Fomitopsis officinalis and Trametes versicolor (FoTv), to treat COVID-19-positive outpatients with mild-to-moderate symptoms assigned to self-quarantined and home management. The study aims to establish the safety and feasibility of the use of FoTv vs placebo in 66 total subjects.

DETAILED DESCRIPTION:
Despite biomedical advances, medical intervention for COVID-19 is largely limited to vaccinations and supportive care during the later stages of disease. While antiviral, anti-inflammatory, and antimalarial options have been explored for later stages of disease, fewer studies have been conducted on medications to reduce the risk of outpatient cases progressing to severe disease. Therefore, it is important that we broaden the search to include agents outside of our usual pharmacopeia. Integrative Medicine offers several promising therapeutics that are available today and warrant investigation.

Some of the botanicals used for their possible immune modulating functions include polypore mushrooms. Among these, Turkey Tail (Trametes versicolor) has a long history of use for its immune supporting properties. An RCT examining the effects of Trametes versicolor in breast cancer patients detected increases in lymphocyte counts and natural killer cell functional activity (Torkelson et al, 2012 and Benson et al, 2019) both of which are key to host COVID-19 response. Further investigations into other relevant mushroom species demonstrated that Agarikon (Fomitopsis officinalis) can strongly induce an array of differential cytokine responses associated with both immune-activation and resolution of host defense- induced inflammatory reactions (unpublished). This homeostatic effect deserves attention for COVID-19 given the high mortality rate associated with cytokine storm.

This is a multi-center, randomized, double blind, placebo-controlled clinical trial to evaluate two polypore mushrooms, Fomitopsis officinalis and Trametes versicolor (FoTv), to treat COVID-19-positive outpatients with mild-to-moderate symptoms assigned to self-quarantined and home management. This study aims to establish the safety and feasibility of the use of FoTv vs placebo in 66 total subjects. Subsequent trials will evaluate Chinese herbal medicine as well as the efficacy of FoTv in a larger study population.

ELIGIBILITY:
Inclusion Criteria:

* Positive COVID-19 diagnosis within the prior 72 hours
* Age 18 years and older
* Women of childbearing potential must have a negative urine or serum hCG. Women of childbearing potential must have a negative serum pregnancy test at screening and agree to use contraception throughout the study period.
* Capable of documenting vitals, symptoms, and study product intake daily and communicating this information to the study team
* Willing to avoid alcohol, cannabis, and dairy products during the study period.

Exclusion Criteria:

* Any of the following symptoms which, according to the CDC, require hospitalization:

  1. Trouble breathing
  2. Persistent pain or pressure in the chest
  3. New confusion or inability to arouse
  4. Bluish lips or face
* Current use of investigational agents to prevent or treat COVID-19
* Known liver disease (ALT/AST >3x ULN or diagnosis of cirrhosis)
* Known renal disease (eGFR < 60 ml/min) or acute nephritis.
* Uncontrolled hypertension (SBP>140 or DBP>90 while on medications)
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Shubov, MD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - University of California, Los Angeles, Los Angeles, California
  - University of California, San Diego, San Diego, California

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mushrooms | Placebo
Started | 28 | 26
Completed | 28 | 25
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mushrooms | Placebo | Total
Number analyzed (Participants) | 26 | 24 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.27 (11.098) | 47.71 (17.269) | 45.40 (14.417)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 10 | 8 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 6 | 13
  Not Hispanic or Latino | 19 | 18 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 20 | 22 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 26 | 24 | 50
Total Protein Normal [Count of Participants; unit: Participants] | 22 | 23 | 45
Albumin Normal [Count of Participants; unit: Participants] | 25 | 23 | 48
Alkaline Phosphatase Normal [Count of Participants; unit: Participants] | 24 | 23 | 47
AST Normal [Count of Participants; unit: Participants] — aspartate aminotransferase
  Participants | 25 | 24 | 49
ALT Normal [Count of Participants; unit: Participants] — alanine transaminase
  Participants | 23 | 23 | 46
Total Bilirubin Normal [Count of Participants; unit: Participants] | 26 | 24 | 50
eGFR Normal [Count of Participants; unit: Participants] — estimated glomerular filtration rate
  Participants | 21 | 14 | 35
Prothrombin Time Normal [Count of Participants; unit: Participants] | 24 | 21 | 45
APTT Normal [Count of Participants; unit: Participants] — Activated partial thromboplastin time
  Participants | 22 | 19 | 41
ESR Normal [Count of Participants; unit: Participants] | 20 | 15 | 35
CRP Normal [Count of Participants; unit: Participants] — C-Reactive Protein
  Participants | 13 | 15 | 28
LDH Normal [Count of Participants; unit: Participants] — Lactate dehydrogenase
  Participants | 13 | 9 | 22

OUTCOME MEASURES:

1. Primary Outcome: Total Protein Normal to Abnormal Transition
Description: We examined participants who were normal at Baseline (Day 1). The Normal to Abnormal proportion reflects the proportion of participants with normal values at Day 1 that became abnormal at Day 14 relative to all participants with normal values at baseline.
Time Frame: 14 days
Population: All participants who were normal at baseline were also normal at day 14, so Chi-square statistic could not be computed.
Measure: Number; unit: percentage of participants
Arm/Group | Mushrooms | Placebo
Number analyzed (Participants) | 22 | 23
percentage of participants | 0 | 0

2. Primary Outcome: Albumin Normal to Abnormal Transition
Description: as for outcome 1
Time Frame: 14 days
Measure: Number; unit: percentage of participants
Arm/Group | Mushrooms | Placebo
Number analyzed (Participants) | 25 | 23
percentage of participants | 4 | 0
Statistical Analysis 1: Comparison: Mushrooms vs Placebo; Test type: Other; p = 1.000, Chi-squared, Corrected; ratio of frequencies = .940

3. Primary Outcome: Alkaline Phosphatase Normal to Abnormal Transition
Description: as for outcome 1
Time Frame: 14 days
Population: Chi-square statistic could not be computed because all participants who were normal at baseline were also normal at day 14.
Measure: Number; unit: percentage of participants
Arm/Group | Mushrooms | Placebo
Number analyzed (Participants) | 24 | 23
percentage of participants | 0 | 0

4. Primary Outcome: AST Normal to Abnormal Transition
Description: as for outcome 1
Time Frame: 14 days
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Mushrooms | Placebo
Number analyzed (Participants) | 25 | 24
percentage of participants | 0 | 0

5. Primary Outcome: ALT Normal to Abnormal Transition
Description: as for outcome 1
Time Frame: 14 days
Measure: Number; unit: percentage of participants
Arm/Group | Mushrooms | Placebo
Number analyzed (Participants) | 23 | 23
percentage of participants | 4.3 | 0
Statistical Analysis 1: Comparison: Mushrooms vs Placebo; Test type: Other; p = 1.000, Chi-squared, Corrected; ratio of frequencies = 1.022

6. Primary Outcome: Bilirubin Normal to Abnormal Transition
Description: as for outcome 1
Time Frame: 14 days
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Mushrooms | Placebo
Number analyzed (Participants) | 26 | 24
percentage of participants | 0 | 0

7. Primary Outcome: Adj. EGFR Normal to Abnormal Transition
Description: as for outcome 1
Time Frame: 14 days
Measure: Number; unit: percentage of participants
Arm/Group | Mushrooms | Placebo
Number analyzed (Participants) | 21 | 14
percentage of participants | 28.6 | 0
Statistical Analysis 1: Comparison: Mushrooms vs Placebo; Test type: Other; p = 0.061, Chi-squared, Corrected; ratio of frequencies = 4.828

8. Primary Outcome: Prothrombin Time Normal to Abnormal Transition
Description: as for outcome 1
Time Frame: 14 days
Measure: Number; unit: percentage of participants
Arm/Group | Mushrooms | Placebo
Number analyzed (Participants) | 23 | 21
percentage of participants | 0 | 14.3
Statistical Analysis 1: Comparison: Mushrooms vs Placebo; Test type: Other; p = .100, Chi-squared, Corrected; ratio of frequencies = 3.526

9. Primary Outcome: APTT Normal to Abnormal Transition
Description: as for outcome 1
Time Frame: 14 days
Measure: Number; unit: percentage of participants
Arm/Group | Mushrooms | Placebo
Number analyzed (Participants) | 22 | 20
percentage of participants | 4.5 | 5.0
Statistical Analysis 1: Comparison: Mushrooms vs Placebo; Test type: Other; p = 1.000, Chi-squared, Corrected; ratio of frequencies = .005

10. Primary Outcome: ESR Normal to Abnormal Transition
Description: as for outcome 1
Time Frame: 14 days
Measure: Number; unit: percentage of participants
Arm/Group | Mushrooms | Placebo
Number analyzed (Participants) | 20 | 14
percentage of participants | 0 | 14.3
Statistical Analysis 1: Comparison: Mushrooms vs Placebo; Test type: Other; p = .162, Chi-squared, Corrected; ratio of frequencies = 3.036

11. Primary Outcome: CRP Normal to Abnormal Transition
Description: as for outcome 1
Time Frame: 14 days
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Mushrooms | Placebo
Number analyzed (Participants) | 13 | 14
percentage of participants | 0 | 0

12. Primary Outcome: LDH Normal to Abnormal Transition
Description: as for outcome 1
Time Frame: 14 days
Measure: Number; unit: percentage of participants
Arm/Group | Mushrooms | Placebo
Number analyzed (Participants) | 13 | 8
percentage of participants | 46.2 | 37.5
Statistical Analysis 1: Comparison: Mushrooms vs Placebo; Test type: Other; p = 1.00, Chi-squared, Corrected; ratio of frequencies = .151

13. Secondary Outcome: Total Bilirubin
Description: comparison of the Total Bilirubin of baseline laboratory data with end-of-treatment labs
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Mushrooms | Placebo
Number analyzed (Participants) | 26 | 24
mg/dL
  Baseline | 0.4215 (0.19164) | 0.3650 (0.13197)
  Day 14 | 0.5469 (0.24245) | 0.4216 (0.18950)
Statistical Analysis 1: Comparison: Mushrooms vs Placebo; Test type: Superiority; p = .174, Mixed Models Analysis; F value = 1.908 — Group by Day interaction

14. Secondary Outcome: Prothrombin Time
Description: comparison of the prothrombin time of baseline laboratory data with end-of-treatment labs
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | Mushrooms | Placebo
Number analyzed (Participants) | 26 | 23
sec
  Baseline | 11.515 (0.7656) | 11.448 (0.9258)
  Day 14 | 11.342 (0.5687) | 11.342 (1.1477)
Statistical Analysis 1: Comparison: Mushrooms vs Placebo; Test type: Superiority; p = .846, Mixed Models Analysis; F value = .038 — Group by Day interaction

15. Secondary Outcome: Aspartate Aminotransferase (AST)
Description: Comparison of the aspartate transaminase of baseline laboratory data with end-of-treatment labs
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Mushrooms | Placebo
Number analyzed (Participants) | 26 | 24
U/L
  Baseline | 23.50 (7.814) | 22.92 (6.406)
  Day 14 | 20.73 (4.944) | 20.54 (4.403)
Statistical Analysis 1: Comparison: Mushrooms vs Placebo; Test type: Superiority; p = .841, Mixed Models Analysis; F value = .041 — Day by Group interaction

16. Secondary Outcome: Alanine Transaminase (ALT)
Description: The safety of the study medication will also assessed by a comparison of the alanine transaminase of baseline laboratory data with end-of-treatment labs or on hospital admission labs (for hospitalized patients)
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Mushrooms | Placebo
Number analyzed (Participants) | 26 | 24
U/L
  Baseline | 28.15 (21.780) | 22.92 (10.902)
  Day 14 | 22.62 (11.876) | 19.79 (7.163)
Statistical Analysis 1: Comparison: Mushrooms vs Placebo; Test type: Superiority; p = 0.612, Mixed Models Analysis; F value = 0.261 — day by group interaction

17. Secondary Outcome: Albumin
Description: comparing Albumin of baseline laboratory data with end-of-treatment labs
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Mushrooms | Placebo
Number analyzed (Participants) | 26 | 24
U/L
  Baseline | 4.565 (0.3610) | 4.517 (0.2729)
  Day 14 | 4.638 (0.2899) | 4.558 (0.2933)
Statistical Analysis 1: Comparison: Mushrooms vs Placebo; Test type: Superiority; p = .690, Mixed Models Analysis; F value = .161 — Group by Day interaction

18. Secondary Outcome: Alkaline Phosphatase
Description: comparing the Alkaline Phosphatase of baseline laboratory data with end-of-treatment labs
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Mushrooms | Placebo
Number analyzed (Participants) | 25 | 24
U/L
  Baseline | 75.64 (38.583) | 76.29 (22.894)
  Day 14 | 68.50 (20.090) | 77.54 (19.797)
Statistical Analysis 1: Comparison: Mushrooms vs Placebo; Test type: Superiority; p = 0.109, Mixed Models Analysis; F value = 2.671 — day by group interaction

19. Secondary Outcome: Lactate Dehydrogenase
Description: A secondary exploratory objective will be to evaluate COVID-19 severity among subjects in each of the two medication arms, compared with placebo, as ascertained by comparing the serum Lactate Dehydrogenase level of baseline laboratory data with end-of-treatment labs or on hospital admission labs (for hospitalized patients).
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Mushrooms | Placebo
Number analyzed (Participants) | 26 | 24
U/L
  Baseline | 186.08 (29.020) | 195.38 (41.484)
  Day 14 | 195.77 (33.448) | 207.70 (37.920)
Statistical Analysis 1: Comparison: Mushrooms vs Placebo; Test type: Superiority; p = 0.844, Mixed Models Analysis; F value = 0.039 — day by group interaction

20. Secondary Outcome: C-Reactive Protein
Description: A secondary exploratory objective will be to evaluate COVID-19 severity among subjects in each of the two medication arms, compared with placebo, as ascertained by comparing the serum C-Reactive Protein level of baseline laboratory data with end-of-treatment labs or on hospital admission labs (for hospitalized patients).
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Mushrooms | Placebo
Number analyzed (Participants) | 26 | 24
mg/dL
  Baseline | 0.9437 (1.15630) | 0.5452 (0.38384)
  Day 14 | 0.3325 (0.47883) | 0.3686 (0.44187)
Statistical Analysis 1: Comparison: Mushrooms vs Placebo; Test type: Superiority; p = 0.044, Mixed Models Analysis; F value = 4.280 — day by group interaction

21. Secondary Outcome: Mid-turbinate SARS CoV-2 Viral Load
Description: A secondary exploratory objective will be to evaluate COVID-19 severity among subjects in each of the two medication arms, compared with placebo, as ascertained by changes in the SARS CoV-2 viral loads among mid-turbinate nasal swabs taken on days 0, 4, 7 and 14.
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: copies per mL
Arm/Group | Mushrooms | Placebo
Number analyzed (Participants) | 23 | 21
copies per mL
  Baseline | 15.2895 (4.93549) | 14.9429 (4.65693)
  Day 7 | 27.7164 (9.02866) | 32.3462 (7.83317)
  Day 14 | 37.7235 (5.14676) | 37.4067 (4.78418)
Statistical Analysis 1: Comparison: Mushrooms vs Placebo; Test type: Superiority; p = .989, Mixed Models Analysis; F value = 0.001 — Day by Group interaction

22. Secondary Outcome: Adj. EGFR
Description: A secondary exploratory objective will be to evaluate COVID-19 severity among subjects in each of the two medication arms, compared with placebo, as ascertained by comparing the Adj. EGFR of baseline laboratory data with end-of-treatment labs or on hospital admission labs (for hospitalized patients).
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Mushrooms | Placebo
Number analyzed (Participants) | 23 | 24
mL/min
  Baseline | 111.93848626354 (20.474674486202) | 101.72611717162 (22.886437908934)
  Day 14 | 104.27777159545 (20.422794275258) | 103.86989833636 (21.260168489030)
Statistical Analysis 1: Comparison: Mushrooms vs Placebo; Test type: Superiority; p = 0.010, Mixed Models Analysis; F value = 7.186 — day by group interaction

23. Secondary Outcome: APTT
Description: A secondary exploratory objective will be to evaluate COVID-19 severity among subjects in each of the two medication arms, compared with placebo, as ascertained by comparing the APTT of baseline laboratory data with end-of-treatment labs or on hospital admission labs (for hospitalized patients).
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | Mushrooms | Placebo
Number analyzed (Participants) | 26 | 24
sec
  Baseline | 32.377 (3.0971) | 32.233 (2.9762)
  Day 14 | 32.108 (2.8652) | 31.513 (3.0824)
Statistical Analysis 1: Comparison: Mushrooms vs Placebo; Test type: Superiority; p = .560, Mixed Models Analysis; F value = .345 — Group by Day interaction

24. Secondary Outcome: INR
Description: A secondary exploratory objective will be to evaluate COVID-19 severity among subjects in each of the two medication arms, compared with placebo, as ascertained by comparing the INR of baseline laboratory data with end-of-treatment labs or on hospital admission labs (for hospitalized patients). The INR is a result of a blood test that measures how long it takes for blood to clot, also known as the prothrombin time (PT). The INR is calculated by comparing the PT to the mean normal prothrombin time (MNPT).
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Mushrooms | Placebo
Number analyzed (Participants) | 26 | 23
ratio
  Baseline | 1.073 (0.0604) | 1.048 (0.0593)
  Day 14 | 1.054 (0.0588) | 1.033 (0.0565)
Statistical Analysis 1: Comparison: Mushrooms vs Placebo; Test type: Superiority; p = 0.707, Mixed Models Analysis; F value = 0.143 — day by group interaction

25. Secondary Outcome: ESR
Description: A secondary exploratory objective will be to evaluate COVID-19 severity among subjects in each of the two medication arms, compared with placebo, as ascertained by comparing the ESR of baseline laboratory data with end-of-treatment labs or on hospital admission labs (for hospitalized patients).
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Mushrooms | Placebo
Number analyzed (Participants) | 24 | 19
mm/hr
  Baseline | 12.54 (9.288) | 14.89 (13.780)
  Day 14 | 11.13 (13.766) | 12.68 (10.409)
Statistical Analysis 1: Comparison: Mushrooms vs Placebo; Test type: Superiority; p = 0.765, Mixed Models Analysis; F value = 0.090 — Day by Group interaction

26. Secondary Outcome: Symptom Count
Description: Symptom severity was assessed via a daily questionnaire across Days 0-14, where participants rated their symptoms on a scale of 0 (none or absent) to 3 (severe). A composite measure was created for each day, based on the 12 symptoms most commonly associated with COVID-19 (fever, fatigue, muscle aches, shortness of breath, shortness of breath upon exertion, cough, sore throat, stuffy nose, runny nose, loss of taste, loss of smell, headache), and counting the total number of symptoms present. scores of 1 or more were considered to be present.
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: Total Number of Symptoms
Arm/Group | Mushrooms | Placebo
Number analyzed (Participants) | 26 | 24
Total Number of Symptoms
  Baseline (Day 0) | 7.2308 (2.30318) | 6.8750 (1.98500)
  Day 1 | 6.2692 (2.50691) | 6.7083 (2.49311)
  Day 2 | 5.6154 (2.36773) | 6.1667 (2.86913)
  Day 3 | 4.9615 (2.76378) | 5.7083 (2.83578)
  Day 4 | 3.8077 (2.41693) | 5.2500 (2.95252)
  Day 5 | 3.5385 (2.24910) | 5.0000 (3.20326)
  Day 6 | 3.5000 (2.21359) | 4.5417 (2.57039)
  Day 7 | 3.1538 (2.27495) | 4.1667 (2.68112)
  Day 8 | 2.8077 (2.28069) | 3.6250 (2.85615)
  Day 9 | 2.4615 (2.12096) | 3.1667 (2.64849)
  Day 10 | 2.3077 (2.27630) | 3.0833 (2.68517)
  Day 11 | 1.6923 (2.07402) | 2.7917 (2.81269)
  Day 12 | 1.3077 (1.56893) | 2.6522 (2.26853)
  Day 13 | 1.1538 (1.48842) | 2.3750 (2.42832)
  Day 14 | 1.1154 (1.65715) | 2.1667 (2.23931)
Statistical Analysis 1: Comparison: Mushrooms vs Placebo; Test type: Superiority; p = 0.005, Mixed Models Analysis; F value = 7.835 — day by group interaction

27. Secondary Outcome: Symptom Severities
Description: Symptom severity was assessed via a daily questionnaire across Days 0-14, where participants rated their symptoms on a scale of 0 (none or absent) to 3 (severe). A composite measure was created for each day, based on the 12 symptoms most commonly associated with COVID-19 (fever, fatigue, muscle aches, shortness of breath, shortness of breath upon exertion, cough, sore throat, stuffy nose, runny nose, loss of taste, loss of smell, headache), and summing the total symptom severities. Higher symptom severities indicates a worse outcome. The minimum and maximum were: 0 to 36, respectively.
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mushrooms | Placebo
Number analyzed (Participants) | 26 | 24
units on a scale
  Baseline (Day 0) | 13.6538 (6.62687) | 11.0833 (4.26224)
  Day 1 | 10.4615 (5.57301) | 10.4167 (5.53186)
  Day 2 | 8.8077 (4.63050) | 9.1667 (5.18079)
  Day 3 | 7.2692 (4.17188) | 8.8333 (5.44272)
  Day 4 | 6.0000 (4.40000) | 8.4583 (5.94159)
  Day 5 | 5.6538 (4.36296) | 7.2917 (5.08604)
  Day 6 | 5.7308 (4.26669) | 7.3750 (5.37152)
  Day 7 | 4.8462 (3.94657) | 6.4167 (5.03826)
  Day 8 | 4.1154 (3.65871) | 5.1667 (4.54606)
  Day 9 | 3.8462 (3.71691) | 4.1250 (3.53015)
  Day 10 | 3.4231 (3.63509) | 3.8750 (3.46802)
  Day 11 | 2.4615 (3.03619) | 3.7083 (4.01605)
  Day 12 | 2.1538 (3.19615) | 3.5652 (3.34156)
  Day 13 | 1.9615 (2.77821) | 3.2500 (3.74456)
  Day 14 | 1.6154 (2.65446) | 2.9167 (3.53758)
Statistical Analysis 1: Comparison: Mushrooms vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; F value = 16.56 — day by group interaction

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | Mushrooms | Placebo
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/24
Other Adverse Events (participants affected / at risk) | 1/26 | 2/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mushrooms (N=26) | Placebo (N=24)
high blood pressure (Vascular disorders) | 1 (12) | 1 (2) — an individual with hypertension reported abnormal blood pressure on days 2-6 and 8-14
High Glucose (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — high glulcose level reported in a participant who had diabetes

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-13): https://cdn.clinicaltrials.gov/large-docs/47/NCT04667247/Prot_SAP_003.pdf